CLINICAL TRIAL: NCT06495840
Title: Postoperative Anxiety and Depression Among Older Chinese Patients: a Prospective Observational Study Based on a Multi-center Perioperative Database in China
Brief Title: Postoperative Anxiety and Depression Among Older Chinese Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Peking University First Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Xiangya Hospital of Central South University (Other); Beijing Anzhen Hospital (Other); Central South University (Other); Peking University People's Hospital (Other); Zhejiang University (Other); Fudan University (Other); Sun Yat-sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); China-Japan Friendship Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Taihe Hospital (Other); Zhejiang Provincial People's Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-AD-Prevalence
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-07

CONDITIONS: Depression; Anxiety; Elderly Patients; Non-cardiac Surgery
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elderly patients: elderly patients undergo non-cardiac surgery (aged ≥ 65 years)
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
A multicenter, prospective observational study to describe the socioeconomic characteristics and the occurrence of postoperative anxiety and depression in the Chinese old population.

DETAILED DESCRIPTION:
As China's population ages, the proportion of elderly people undergoing surgery increases. Perioperative anxiety and depression, particularly in elderly patients, is common and associated with multiple medical and social adversities. Previous studies have found a 31 percent risk of anxiety and 29 percent risk of depression in older perioperative patients. However, nationally representative epidemiological data for postoperative anxiety and depression, in particular elderly patients undergoing non-cardiac surgery, are unavailable in China. Therefore, providing nationwide epidemiological data on postoperative anxiety and depression in Chinese elderly patients provides a valuable opportunity for policy makers and health care professionals to optimize the management of geriatric mental health in China.

ELIGIBILITY:
Inclusion Criteria:

1. elderly patients (age ≥ 65 years)
2. undergoing elective surgery with a planned overnight hospital stay following surgery
3. non-cardiac surgery, non-neurosurgical surgery

Exclusion Criteria:

1. patients fully refused to participate in the study
2. patients with severe dementia, language disorder, severe hearing or visual impairment, coma, and end-stage status
3. patients whose surgeries were canceled
4. history of previous severe mental illness or long-term use of psychotropic medications
5. patients admitted to ICU immediately after surgery
6. patients who died within 7 days after surgery
7. patients who did not complete the scale assessment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (aged ≥ 65 years) who completed the anxiety and depression assessment after the elective noncardiac, non-neurosurgical surgery were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 8590 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Anxiety | within 7 days after surgery
  The GAD-7 is a seven-item questionnaire for screening on the presence of generalized anxiety disorder and assessing its severity. Items were scored on a four-point scale with total scores ranging from zero to twenty-one. Scores were defined as: ≥5 mild, ≥10 moderate, and ≥15 severe anxiety. The recommended screening cutoff was ≥10, corresponding with at least a moderate level of anxiety. Higher scores mean more anxiety.
Depression | within 7 days after surgery
  Primary outcomes were depression Patient Health Questionnaire 9 (PHQ-9).The PHQ-9 is a nine-item questionnaire for screening on the presence of depressive symptoms and monitoring depression severity. Items were scored on a four-point scale with total scores ranging from zero to twenty-seven. Scores were defined as: ≥5 mild, ≥10 moderate, and ≥15 severe level of depression. The recommended screening cutoff was ≥10, corresponding with at least a moderate level of depression. The higher the score, the worse the situation. The total score ranges from 0 to 27, and higher scores indicate more depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- First Medical center of Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided